CLINICAL TRIAL: NCT02978495
Title: Neoadjuvant Carboplatin in Triple Negative Breast Cancer - A Prospective Phase II Study (NACATRINE Trial).
Brief Title: Neoadjuvant Carboplatin in Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Cristiano de Padua, Principal Investigator, Barretos Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BarretosCH - 20162
Record Dates: First submitted 2016-11-24; First posted 2016-12-01 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: BRCA1 Hereditary Breast and Ovarian Cancer Syndrome
MeSH Terms: interventions — Doxorubicin; Carboplatin; Paclitaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A- BRCA Mutation (Experimental): 1. Doxorrubicin 60 mg/m2 concomitantly with Cyclophosphamide 600mg/m2, every 3 weeks, for 4 cycles followed by:
  2. Paclitaxel 80 mg/m2 once a week, for 12 weeks, concomitant to Carboplatin AUC 1,5 once a week, for 12 weeks.
  Interventions: Drug: Doxorubicin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Cyclophosphamide
- B- BRCA Mutation (Active Comparator): 1. Doxorrubicin 60 mg/m2 concomitantly with Cyclophosphamide 600mg/m2, every 3 weeks, for 4 cycles followed by:
  2. Paclitaxel 80 mg/m2 once a week, for 12 weeks.
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel; Drug: Cyclophosphamide
- C- BRCA wild-type (Experimental): 1. Doxorrubicin 60 mg/m2 concomitantly with Cyclophosphamide 600mg/m2, every 3 weeks, for 4 cycles followed by:
  2. Paclitaxel 80 mg/m2 once a week, for 12 weeks, concomitant to Carboplatin AUC 1,5 once a week, for 12 weeks.
  Interventions: Drug: Doxorubicin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Cyclophosphamide
- D- BRCA wild-type (Active Comparator): 1. Doxorrubicin 60 mg/m2 concomitantly with Cyclophosphamide 600mg/m2, every 3 weeks, for 4 cycles followed by:
  2. Paclitaxel 80 mg/m2 once a week, for 12 weeks.
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Doxorubicin — Doxorrubicin 60 mg/m2 4 cycles each 21 days
Drug: Carboplatin — Carboplatin AUC 1,5 once a week, for 12 weeks
  Arms: A- BRCA Mutation; C- BRCA wild-type
Drug: Paclitaxel — 80mg/m2 weekly for 12 weeks
Drug: Cyclophosphamide — 600mg/m2 4 cycles each 21 days

SUMMARY:
Breast cancer is the most frequent neoplasm in women in Brazil and in the world and up to 15% of all cases diagnosed correspond to the triple negative subtype. Triple negative breast cancer affects young women with germline mutations in BRCA 1/2 genes. Giving the lack of target therapies to date, there is no consensus regarding the most effective treatment for this subgroup of tumors. Although evidence shows that triple negative breast cancer is highly sensitive to chemotherapy when compared to other breast tumors, there is no evidence to support the hypothesis that patients with triple negative breast cancer and mutation in BRCA1 / 2 genes have higher chemosensitivity to neoadjuvant therapy. The investigator proposes a prospective, randomized, open-label, phase II study, evaluating the rate of complete pathologic response, disease-free survival, overall survival and prognostic evaluation of BRCA1 / 2 mutation status in women with triple negative breast cancer submitted to sequential neoadjuvant chemotherapy based on anthracycline and taxane, with or without carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Triple Negative Breast Cancer;
* Stage II or III;
* Performance Status ECOG <2 or Karnofsky >50%;
* Hematologic (minimal values):

Absolute neutrophil count > 1,500/mm3 Hemoglobin > 10.0 g/dl Platelet count > 100,000/mm3

Exclusion Criteria:

* Stage I or IV;
* other malignancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR), defined as absence of invasive cancer in the breast and axillary lymph nodes. | within the first 21 days after surgery

SECONDARY OUTCOMES:
Disease free survival (DFS) | within the first 60 month after surgery
Overall survival (OS) | within the first 60 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] von Minckwitz G, Schneeweiss A, Loibl S, Salat C, Denkert C, Rezai M, Blohmer JU, Jackisch C, Paepke S, Gerber B, Zahm DM, Kummel S, Eidtmann H, Klare P, Huober J, Costa S, Tesch H, Hanusch C, Hilfrich J, Khandan F, Fasching PA, Sinn BV, Engels K, Mehta K, Nekljudova V, Untch M. Neoadjuvant carboplatin in patients with triple-negative and HER2-positive early breast cancer (GeparSixto; GBG 66): a randomised phase 2 trial. Lancet Oncol. 2014 Jun;15(7):747-56. doi: 10.1016/S1470-2045(14)70160-3. Epub 2014 Apr 30. PMID 24794243
- [Result] Gerber B, Loibl S, Eidtmann H, Rezai M, Fasching PA, Tesch H, Eggemann H, Schrader I, Kittel K, Hanusch C, Kreienberg R, Solbach C, Jackisch C, Kunz G, Blohmer JU, Huober J, Hauschild M, Nekljudova V, Untch M, von Minckwitz G; German Breast Group Investigators. Neoadjuvant bevacizumab and anthracycline-taxane-based chemotherapy in 678 triple-negative primary breast cancers; results from the geparquinto study (GBG 44). Ann Oncol. 2013 Dec;24(12):2978-84. doi: 10.1093/annonc/mdt361. Epub 2013 Oct 17. PMID 24136883
- [Result] Byrski T, Gronwald J, Huzarski T, Grzybowska E, Budryk M, Stawicka M, Mierzwa T, Szwiec M, Wisniowski R, Siolek M, Dent R, Lubinski J, Narod S. Pathologic complete response rates in young women with BRCA1-positive breast cancers after neoadjuvant chemotherapy. J Clin Oncol. 2010 Jan 20;28(3):375-9. doi: 10.1200/JCO.2008.20.7019. Epub 2009 Dec 14. PMID 20008645
- [Result] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Result] Valsecchi ME, Kimmey G, Bir A, Silbermins D. Role of Carboplatin in the Treatment of Triple Negative Early- Stage Breast Cancer. Rev Recent Clin Trials. 2015;10(2):101-10. doi: 10.2174/1574887110666150624101343. PMID 26104428
- [Result] Arun B, Bayraktar S, Liu DD, Gutierrez Barrera AM, Atchley D, Pusztai L, Litton JK, Valero V, Meric-Bernstam F, Hortobagyi GN, Albarracin C. Response to neoadjuvant systemic therapy for breast cancer in BRCA mutation carriers and noncarriers: a single-institution experience. J Clin Oncol. 2011 Oct 1;29(28):3739-46. doi: 10.1200/JCO.2011.35.2682. Epub 2011 Sep 6. PMID 21900106
- [Result] Gonzalez-Angulo AM, Timms KM, Liu S, Chen H, Litton JK, Potter J, Lanchbury JS, Stemke-Hale K, Hennessy BT, Arun BK, Hortobagyi GN, Do KA, Mills GB, Meric-Bernstam F. Incidence and outcome of BRCA mutations in unselected patients with triple receptor-negative breast cancer. Clin Cancer Res. 2011 Mar 1;17(5):1082-9. doi: 10.1158/1078-0432.CCR-10-2560. Epub 2011 Jan 13. PMID 21233401
- [Result] Paluch-Shimon S, Friedman E, Berger R, Papa M, Dadiani M, Friedman N, Shabtai M, Zippel D, Gutman M, Golan T, Yosepovich A, Catane R, Modiano T, Kaufman B. Neo-adjuvant doxorubicin and cyclophosphamide followed by paclitaxel in triple-negative breast cancer among BRCA1 mutation carriers and non-carriers. Breast Cancer Res Treat. 2016 May;157(1):157-65. doi: 10.1007/s10549-016-3800-5. Epub 2016 Apr 25. PMID 27113739
- [Result] Muendlein A, Rohde BH, Gasser K, Haid A, Rauch S, Kinz E, Drexel H, Hofmann W, Schindler V, Kapoor R, Decker T, Lang AH. Evaluation of BRCA1/2 mutational status among German and Austrian women with triple-negative breast cancer. J Cancer Res Clin Oncol. 2015 Nov;141(11):2005-12. doi: 10.1007/s00432-015-1986-2. Epub 2015 May 15. PMID 25971625